CLINICAL TRIAL: NCT02635503
Title: A Prospective Randomized Controlled Trial Comparing Totally Laparoscopic Resection With Natural Orifice Specimen Extraction (NOSE) Versus Conventional Laparoscopic Surgery for Sigmoid Colon or Rectal Cancer
Brief Title: Safety Study of Totally Laparoscopic Resection With Natural Orifice Specimen Extraction (NOSE) for Rectosigmoid Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zhixiang Zhou, director of Colorectal surgical Department, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC2015SF-04
Record Dates: First submitted 2015-11-30; First posted 2015-12-21 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; laparoscopic surgery; natural orifice specimen extraction; Inflammatory response
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- transrectal specimen extraction (Experimental): Laparoscopic colorectal resection with natural orifice specimen extraction will be performed for patients in this group.
  Interventions: Procedure: transrectal specimen extraction
- Conventional laparoscopic surgery (Active Comparator): Conventional laparoscopic surgery for colorectal cancer will be performed for patients in this group.
  Interventions: Procedure: Conventional laparoscopic surgery

INTERVENTIONS:
Procedure: transrectal specimen extraction — After mobilization of bowel and dissection of lymph nodes, a cross clamp was placed distal to the tumor. Distal rectum was transected after fully disinfecting rectal lumen by 10% povidone-iodine. An anvil head attached to circular stapling device was put into abdominal cavity through rectal stump, and put into colon lumen through a longitudinal incision, then the proximal colon was transected in close proximity to the upper pole of incision by a linear stapling device. During specimen extraction though the rectum, a disposable sterile protective cover was used to avoid cancer cell exfoliation and implantation. The rectal opening was reclosed by a linear stapler. End-to-end colorectal anastomosis was performed with a circular stapler using the double-stapling technique.
  Other Names: NOSE
  Arms: transrectal specimen extraction
Procedure: Conventional laparoscopic surgery — High ligation of inferior mesenteric vessel , mobilization of bowel, and dissection of lymph nodes were performed laparoscopically, and total mesorectal excision with nerve-sparing technique was followed for rectal cancer. Conventional laparoscopic-assisted surgery (CLS), a small incision with a 3-7cm length was made in hypogastrium, transection of rectum was completed through abdominal incision, then the specimen was removed and the bowel was prepared for anastomosis. The anastomosis for all rectal cancer and most of sigmoid colon cancer was performed by a double-stapling technique following open resection.
  Other Names: CLS
  Arms: Conventional laparoscopic surgery

SUMMARY:
The purpose of this study is to compare the safety and efficacy of laparoscopic resection with natural orifice specimen extraction versus conventional laparoscopic surgery for sigmoid colon or rectal cancer.

DETAILED DESCRIPTION:
Further study details as provided by Chinese Academy of Medical Sciences.

ELIGIBILITY:
Inclusion Criteria:

* 18 years < age < 80 years
* Tumor located in rectosigmoid (defined as 8- to 30-cm from the anal verge)
* Pathological rectosigmoid adenocarcinoma
* Preoperative T stage ranging from T1 to T4a according to the 7th Edition of American Joint Committee on Cancer (AJCC) Staging Manual
* Tumor size of 6 cm or less;
* Eastern Cooperative Oncology Group (ECOG) score is 0-1
* American Society of Anesthesiology (ASA) score is Ⅰ-Ⅲ
* Informed consent

Exclusion Criteria:

* Body mass index (BMI) >30 kg/m2
* Pregnant woman or lactating woman
* Severe mental disease
* Previous abdominal surgery
* Emergency operation due to complication (bleeding, perforation or obstruction) caused by colorectal cancer
* Requirement of simultaneous surgery for other disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2015-11; Primary Completion 2020-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Early morbidity rate | 30 days
  The early morbidity rate is defined as the event observed during operation and within 30 days after surgery.

SECONDARY OUTCOMES:
Duration of the intervention | 1 day
  Duration of surgery.
Peritoneal bacterial contamination | 1 day
  Peritoneal fluid samples were collected under sterile conditions at the end of the procedure and sent for gram stain as well as anaerobic, aerobic, and fungal cultures.We assess the contamination rate of peritoneal fluid in the two interventions.
Pain score | 14 days
  Recording of the needed analgesia guided by pain score
3-year disease free survival rate | 3 years
  A survival analysis will be performed using the Kaplan-Meier method, for which a comparison of the survival curve will also made using a Log-rank test.
5-year overall survival rate | 5 years
  A survival analysis will be performed using the Kaplan-Meier method, for which a comparison of the survival curve will also made using a Log-rank test.
Plasma levels of several cytokines after colorectal cancer surgery | 7 days
  We have measured and compared perioperative plasma levels of interleukin-2, interleukin-6, interleukin-8, C-reactive protein and procalcitonin in the two group sample.

CONTACTS AND LOCATIONS:
Overall Officials: Zhixiang Zhou, M.D., Principal Investigator — Cancer Hospital, Chinese Academy of Medical Sciences, Peking Union Medical College
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No